CLINICAL TRIAL: NCT03212508
Title: Comparison of Two Nasal Interface for Continuous Distending Airway Pressure in Preterm Infants: RAM Nasal Cannula and Hudson Prongs
Brief Title: Comparison of Two Nasal Interface for CPAP in Preterm
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00029410
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: Continuous positive airway pressure, preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: RAM cannula and Hudson prongs — Measuring intraoral pressure using two different nasal interface for applying nasal continuous positive airway pressure

SUMMARY:
Continuous distending airway pressure (CPAP) has gained popularity as a means to provide non-invasive respiratory support in neonates to reduce ventilator induced lung injury (VILI). However, maintaining CPAP in preterm infants has been challenging, often related to issues with nasal interface such as nasal septal injury, problems with keeping the prongs in the nose and leak around the prongs with are important factors in proving effective CPAP. RAM cannula was recently approved for providing supplemental oxygen and soon adapted by many centers to provide CPAP in preterm infants. Concerns have been raised that RAM cannula interface results in sub-optimal pressure delivery compared to standard nasal prongs.

DETAILED DESCRIPTION:
Objective:

To compare efficacy of delivering continuous distending pressure in preterm neonates using RAM cannula versus the standard prongs (Hudson prongs) by measuring intra-oral pressure. It is hypothesize that CPAP delivered with RAM cannula is comparable to pressure delivered via standard nasal interface in routine clinical practice; and the desired CPAP level is often not achieved in presence of variable leak from mouth irrespective of type of nasal interface.

Aim 1: Compare the level of CPAP in oral cavity between RAM cannula and Hudson prong nasal interface in preterm Hypothesis: The intraoral pressure with CPAP will not be different with use of RAM cannula or Hudson prong nasal interface

Aim 2: Evaluate the effect of nasal interface (RAM cannula and Hudson prong) on respiratory variables Hypothesis: There will be no difference in respiratory variables with CPAP delivered by RAM cannula compared to Hudson prongs.

Method:

This was a single center prospective study. Inclusion criteria: Any preterm with respiratory distress requiring CPAP but not mechanical ventilation or NIPPV was eligible for the study. 12 preterm infant more than 48 hours old and stable on bubble CPAP were recruited for the study Exclusion criteria: Infants with major congenital anomalies, neuromuscular disorders, upper airway anomalies, critically sick infants

CPHS approval and parental consent was obtained prior to enrollment in the study.

Each infant was studied for ~1 hour during which the oral pressure was measured while receiving CPAP with RAM nasal cannula interface and then with Hudson prongs. Blinding of the intervention (nasal interface) was not feasible because of the visible differences in the two nasal interfaces.

Procedure: Intra-oral pressure measured via a differential pressure transducer while infant in receiving CPAP, and digitized data recorded with each nasal interface ( goal to record at least 20 sec of stable waveform on each nasal interface). Standard care provided during the study period and no changes made with CPAP level or flow.

The difference between set pressure and measured pressure with RAM cannula and Hudson prong was compared with standard paired student t-test with 95% confidence limits. Difference in other variables will be similarly compared with t-test. STAT 12 will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Any preterm with respiratory distress requiring CPAP but not mechanical ventilation or NIPPV will be eligible for the study. We will recruit preterm infant more than 48 hours old and stable on bubble CPAP

Exclusion Criteria:

* Infants with major congenital anomalies, neuromuscular disorders, upper airway anomalies, critically sick infants

Ages: 48 Hours to 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any preterm with respiratory distress requiring CPAP
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
The difference between set pressure and measured pressure with RAM cannula and Hudson prong | one hour
  Intraoral pressure measure using a differential pressure transducer with RAM cannula and then with Hudson prongs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh N, McNally MJ, Darnall RA. Does the RAM Cannula Provide Continuous Positive Airway Pressure as Effectively as the Hudson Prongs in Preterm Neonates? Am J Perinatol. 2019 Jul;36(8):849-854. doi: 10.1055/s-0038-1675330. Epub 2018 Nov 5. PMID 30396227